CLINICAL TRIAL: NCT02932969
Title: A Randomized, Double-Blind, Placebo-controlled, Single Continuous Intravenous Infusion Study of BMS-986231 to Assess Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics in Healthy Japanese and Non- Asian Participants
Brief Title: Study With Healthy Japanese and Non-Asian Participants With BMS-986231
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CV013-018
Record Dates: First submitted 2016-10-12; First posted 2016-10-13 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Heart Decompensation, Acute
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Panel 1 Arm (Experimental): BMS-986231 and BMS-986231 Placebo intravenously
  Interventions: Drug: BMS-986231; Drug: BMS-986231 Placebo
- Panel 2 Arm (Experimental): BMS-986231 and BMS-986231 Placebo intravenously
  Interventions: Drug: BMS-986231; Drug: BMS-986231 Placebo
- Panel 3 Arm (Experimental): BMS-986231 and BMS-986231 Placebo intravenously
  Interventions: Drug: BMS-986231; Drug: BMS-986231 Placebo

INTERVENTIONS:
Drug: BMS-986231
Drug: BMS-986231 Placebo

SUMMARY:
The purpose of this Phase 1 study is to evaluate the safety, tolerability, PK, and pharmacodynamics (PD) of BMS-986231 in healthy Japanese and Non-Asian participants. There is no formal hypothesis to be statistically tested.

ELIGIBILITY:
Inclusion Criteria:

* Ancestry

  * First generation Japanese
  * Non-Asian with grandparents and parents of non-Asian descent
* Body weight greater than or equal to 45kg and less than or equal to 110kg
* Women of childbearing potential have specific birthcontrol methods
* Males sexually active with women of childbearing potential have specific birthcontrol methods

Exclusion Criteria:

* History of chronic illness
* Chronic headaches
* Recurrent dizziness
* Personal or family history of heart disease
* Personal history of bleeding diathesis

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2017-05-26 (Actual); Study Completion 2017-05-26 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single continuous IV infusion of BMS-986231 in healthy Japanese and Non-Asian participants based on Adverse events, clinical laboratory values, vital signs, ECGs, and physical examinations | 11 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- West Coast Clinical Trials, Llc, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Education Resource — http://www.bms.com/studyconnect/pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx